CLINICAL TRIAL: NCT03211793
Title: Mesenchymal Stromal Cells for Angiogenesis and Neovascularisation in Digital Ulcers of Systemic Sclerosis: the MANUS Trial
Brief Title: Mesenchymal Stromal Cells as Treatment for Digital Ulcers in Systemic Sclerosis
Acronym: MANUS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, prof dr. M. C. Verhaar, prof. dr., UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MANUS; 2015-000168-32 (EudraCT Number)
Record Dates: First submitted 2017-04-27; First posted 2017-07-07 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Systemic Sclerosis; Digital Ulcer
Keywords: systemic sclerosis; scleroderma; digital ulcer; vasculopathy; mesenchymal stromal cell; mesenchymal stem cell
MeSH Terms: conditions — Scleroderma, Systemic; digital ulcers; Scleroderma, Diffuse; Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MSC injections (Experimental): Intramuscular injection of mesenchymal stromal cells (50 million allogeneic MSCs in 0.9% NaCl and 10% human serum albumin).
  Interventions: Drug: Mesenchymal stromal cells
- Placebo injections (Placebo Comparator): Intramuscular injection of placebo (NaCl 0.9% + 10% human serum albumin)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mesenchymal stromal cells — 8 intramuscular injections at designated sites in the hand/forearm muscles of the most affected side. Blinded syringes will be used. Injections will be administered by an experienced clinician (plastic surgeon or hand surgeon).
  Arms: MSC injections
Other: Placebo — 8 intramuscular injections at designated sites in the hand/forearm muscles of the most affected side. Blinded syringes will be used. Injections will be administered by an experienced clinician (plastic surgeon or hand surgeon).
  Arms: Placebo injections

SUMMARY:
The MANUS Trial aims to examine the safety, feasibility and potential efficacy of intramuscularly injected allogeneic mesenchymal stromal cells as treatment for digital ulcers of systemic sclerosis.

DETAILED DESCRIPTION:
The MANUS Trial is a randomized double-blind, placebo-controlled clinical trial. Patients with systemic sclerosis (SSc) and digital ischemia with intractable ischemic digital ulcers refractory to conventional treatments are eligible to participate.

20 participants will be randomised (1:1) to undergo intramuscular injection (8 sites) of allogeneic bone marrow derived mesenchymal stromal cells (BM-MSC) (45-50*10^6) or placebo in the most affected limb.

Main study parameters/endpoints: The primary outcome is the toxicity of the treatment at 12 weeks after MSC administration, defined as

1. Local toxicity, including signs of local inflammation (swelling, warmth, impairment of function), worsening of ulcers or new ulcers or hematomas after MSC administration
2. Other adverse events, graded according to the Common Terminology Criteria for Adverse Events version 4.0, expressed as maximum grade toxicity per organ system.

Secondary outcome measures are: number of serious adverse events, pain and disability parameters; healing, time to healing and reduction of new ischemic digital ulcers; modified Rodnan skin score; Scleroderma Health Assessment Questionnaire (S-HAQ) including visual analogue scales (VAS) for scleroderma-specific symptoms; Quality-of-life (SF-36, EuroQol (EQ-5D); Cochin hand function score. We will also evaluate changes in capillary morphology and architecture using capillaroscopy; biochemical parameters; markers for endothelial activation and injury, inflammation, oxidative stress, circulating cells including endothelial cells, hematopoietic and endothelial progenitor cells, cytokines and growth factors, immunological responses. Follow-up visits will be scheduled at 48 hours and 2, 4, 8, 12, 24 and 52 weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of SSc according to the 2013 ACR/EULAR criteria
* At least one active digital ulcer (painful area, >2 mm in diameter with visible depth and loss of dermis) refractory to intravenous prostacyclins

  * 'Refractory to prostacyclins' is defined as
  * Worsening of ulcer(s) within 1 month after prostacyclins iv
  * No improvement of ulcer(s) after 2 months after prostacyclins iv, as judged by the referring physician
  * Recurrence of exactly the same ulcer(s) (same location) within 3 months after prostacyclins iv
* Written informed consent

Exclusion Criteria:

* Ulcer with underlying calcinosis (ruled out by X-ray prior to screening/inclusion)
* History of neoplasm or malignancy in the past 10 years
* Pregnancy or unwillingness to use adequate contraception during study
* Serious known concomitant disease with life expectancy <1 year
* Uncontrolled hypertension
* Uncontrolled acute or chronic infection with systemic symptoms (e.g. fever)
* Follow-up impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Toxicity of the treatment | 12 weeks after MSC administration
  Toxicity of the treatment is defined as 1. Local toxicity, including signs of local inflammation (swelling, warmth, impairment of function), worsening of ulcers or new ulcers or hematomas after MSC administration 2. Other adverse events, graded according to the Common Terminology Criteria for Adverse Events version 4.0, expressed as maximum grade toxicity per organ system.

SECONDARY OUTCOMES:
Serious adverse events | 48 hours, 2, 4, 8, 12, 24 weeks and 52 weeks after MSC administration
  Any treatment-related serious adverse events (SAE) defined as events leading to hospitalization, death, or persistent or significant disability. To establish the presence or absence of a causal relationship, the World Health Organisation guidelines for pharmacovigilance will be followed.
Change in perceived pain based on the Numerical Rating Scale | 48 hours, 2, 4, 8, 12, 24 weeks and 52 weeks after MSC administration
  Change in pain as assessed using the Numerical Rating Scale,
Change in perceived pain based on the digital ulcer visual analogue scale (part of the S-HAQ) | 48 hours, 2, 4, 8, 12, 24 weeks and 52 weeks after MSC administration
  Change in pain as assessed using the digital ulcer visual analogue scale (part of the S-HAQ).
Change in perceived pain based on the pain VAS ( part of the S-HAQ) | 48 hours, 2, 4, 8, 12, 24 weeks and 52 weeks after MSC administration
  Change in pain as assessed using the pain VAS (S-HAQ), use of analgesics.
Change in perceived pain based on the use of analgesics. | 48 hours, 2, 4, 8, 12, 24 weeks and 52 weeks after MSC administration
  Change in pain as assessed by analyzing the use of analgesics.
Quality of life - SF-36 | 12, 24 and 52 weeks after MSC administration
  SF-36 questionnaire.
Quality of life - Euroqol | 12, 24 and 52 weeks after MSC administration
  EuroQol questionnaire
Disability | 12, 24 and 52 weeks after MSC administration
  Assessed with the HAQ-DI questionnaire.
Hand function | 12, 24 and 52 weeks after MSC administration
  Cochin Hand Function Score
Number (and change in number) of digital ulcers | 48 hours, 2, 4, 8, 12, 24 weeks and 52 weeks after MSC administration
Healing of digital ulcers | 48 hours, 2, 4, 8, 12, 24 weeks and 52 weeks after MSC administration
  Healing of ulcers is defined as complete epithelialization, regardless of residual pain. This will be established using sequential pictures in addition to the clinical examination.
Ulcer size | 48 hours, 2, 4, 8, 12, 24 weeks and 52 weeks after MSC administration
  Using sequential pictures, ulcer area and circumference will be measured.
Time to healing of digital ulcers | 48 hours, 2, 4, 8, 12, 24 weeks and 52 weeks after MSC administration
Need to alter medication regime | 48 hours, 2, 4, 8, 12, 24 weeks and 52 weeks after MSC administration
  The need to alter the medication regime as determined by the patient's attending rheumatologist.
Modified Rodnan Skin Score | 12, 24 and 52 weeks after MSC administration
Severity of Raynaud's symptoms | 12 , 24 and 52 weeks after MSC administration
  Raynaud Condition Score
Changes in capillary morphology and architecture | 2, 12, 24 weeks and 52 weeks after MSC administration
  as visualized with video-assisted nailfold capillaroscopy by a trained investigator. The images will be scored by a certified rheumatologist and a trained investigator.
Changes in laboratory parameters | 48 hours, 2, 4, 8, 12 weeks after MSC administration
  A range of haematological and chemical parameters will be measured for safety assessment. Additionally, serum, plasma and peripheral blood mononuclear cells will be collected and stored for analysis at a later time point. Samples will be analysed and used to assess markers for endothelial activation and injury, proangiogenic factors, inflammation and oxidative stress. The presence of HLA-antibodies will be determined as well.
Changes in circulating cell populations | 48 hours, 2, 4, 8, 12 weeks after MSC administration
  Circulating cell populations will be studied by immunofluorescence labelling and analysis using fluorescence assisted cell sorting (FACS Canto machine).

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Verhaar, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Rhijn-Brouwer FCC, Gremmels H, Fledderus JO, Schuurman AH, Bonte-Mineur F, Vonk MC, Voskuyl AE, de Vries-Bouwstra JK, Coert JH, Radstake TRDJ, van Laar JM, Verhaar MC; MANUS Study Group. A randomised placebo-controlled double-blind trial to assess the safety of intramuscular administration of allogeneic mesenchymal stromal cells for digital ulcers in systemic sclerosis: the MANUS Trial protocol. BMJ Open. 2018 Aug 20;8(8):e020479. doi: 10.1136/bmjopen-2017-020479. PMID 30127049